CLINICAL TRIAL: NCT04048044
Title: THE EFFECTS OF THE RejuvaMatrix ™ ON TELOMERES
Brief Title: EFFECTS OF RejuvaMatrix ™ ON TELOMERES
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Holos Institutes of Health, Inc (Other)
Responsible Party: Principal Investigator, C. Norman Shealy, M.D., Ph.D., Holos Institutes of Health, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HIH RM
Record Dates: First submitted 2012-05-10; First posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2012-05

CONDITIONS: Telomeres

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Telomere length, GigaHz exposure (Active Comparator): Measurement of white blood cell telomeres before and yearly for 5 years
  Interventions: Device: Exposure to GHz electromagnetic energy (RejuvaMatrix)

INTERVENTIONS:
Device: Exposure to GHz electromagnetic energy (RejuvaMatrix) — 75 decibels of 54 to 78 GHz daily for 60 minutes

SUMMARY:
Lying for 30 to 60 minutes daily in a field of 75 decibels of electromagnetic energy at 54 to 78 GHz will allow telomeres of white blood cells to regenerate

DETAILED DESCRIPTION:
Individuals who are post menopausal and who do not have an implanted electronic device, such as a pacemaker will have base line white blood cell telomeeres measured at Repeat Diagnostics in Vancouver. They will be supplied with a two inch foam mat in the center of which is copper screen with one pound of crushed sapphire. The mat looks like a mattreess and is placed on top of the regular mattress. Participants are provided with a Tesla coil to be attached to a copper wire coming from the copper screen. They will also be provided with a timer so that they can set the Tesla coil to be activated for a maximum of 60 minutes while they sleep.

Telomeres will be measured at the end of each year for 5 years.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Implanted electronic device
* Major, debilitating disease
* Person living with an individual who has an implanted device
* Person who is or could become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Length of telomeres after 5 years compared with baseline | 5 years

SECONDARY OUTCOMES:
Total Symptom Index | 5 years